CLINICAL TRIAL: NCT03875222
Title: Studying New Criteria for Prediction of Site of Accessory Pathway From Surface ECG
Brief Title: New Criteria for Accessory Pathway Localization From Surface ECG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidy Yacoup Daoud Danial, principle investigator, Assiut University
Other Study IDs: Accessory pathway location
Record Dates: First submitted 2019-03-13; First posted 2019-03-14 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Accessory Pathway
MeSH Terms: conditions — Pre-Excitation Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
study for discovering new criteria for localization of site of accessory pathway from surface ECG

DETAILED DESCRIPTION:
the study aims for discovering new criteria for percise localization of accessory pathway from surface ECG in referance to final flouroscopic ablation site

ELIGIBILITY:
Inclusion Criteria:

* any patient with manifest accessory pathway .

Exclusion Criteria:

* multiple accessory pathways .previous ablation.

Ages: 10 Years to 90 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: any patient with manifest accessory pathway between 10 and 90 years of age undergoing EP maping and ablation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
percise localization of accessory pathway from surface ECG in referance to successful ablation site | 2 years
  successful localization of accessory pathway from surface ECG in referance to successful ablation site during EP maping